CLINICAL TRIAL: NCT02218346
Title: A Phase 1, Two-Way Crossover Study to Assess the Pharmacokinetics and Safety of a Single Dose of AG-221 in Healthy Male Subjects When Administered Under Fed and Fasted Conditions
Brief Title: Food Effect Study of AG-221 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG221-C-002
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (unfed) (Active Comparator): Treatment A: Single oral dose of AG-221 mesylate at Hour 0 on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: AG221
- Treatment B (fed) (Active Comparator): Treatment B: Single oral dose of AG-221 mesylate at Hour 0 on Day 1, 30 minutes after the start of a high-fat breakfast.
  Interventions: Drug: AG221

INTERVENTIONS:
Drug: AG221 — AG221 in fed and fasted conditions

SUMMARY:
AG-221 is a first-in-class drug targeted specifically to inhibit the IDH2 enzyme. Small molecule inhibition of the IDH enzyme represents a new, targeted approach to cancer treatment.

Administration of oral drugs with food may change the absorption of drugs, and it is therefore useful to characterize the effect of food early in drug development.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects 18 to 56 years of age, inclusive, at Screening.
2. Subjects who are able to understand and sign informed consent prior to the conduct of any protocol-specific screening procedures.
3. Subjects must be willing and able to complete all study assessments and procedures.
4. Subjects, with the exception of those who have undergone vasectomy at least 6 months prior to Screening, must agree to use condom with spermicide as contraception (regardless of their female partner's childbearing potential or their partner's use of their own contraception) from Day 1 of Period 1 until 28 days following the last dose of study drug.
5. Subjects must have a body weight ≥50 kg and body mass index (BMI) ≥18.5 and ≤32 kg/m2 at Screening.
6. Subjects must be in general good health as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, and 12-lead ECGs at Screening or on Day -1 of each period.
7. Subjects must be non-smokers and have not used nicotine-containing products for at least 3 months prior to Screening.
8. Subjects must be willing to refrain from caffeine- or xanthene-containing products (coffee, tea, cola, chocolate, etc.) for 48 hours prior to dosing in each period and through discharge from the study center.
9. Subjects must be willing to refrain from strenuous exercise starting 72 hours prior to Day 1 of Period 1 through the Follow-up visit.
10. Subjects must be willing to refrain from ingestion of alcohol starting 7 days (14 days for red wine) prior to Day 1 of Period 1 through the Follow-up visit.
11. Subjects must agree not to donate blood or plasma to any blood bank or for any purpose (other than blood samples in this study) for the duration of participation in the study (from Screening to Follow-up).

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled in the study:

1. Subjects who have previously received AG-221 (this does not apply at Period 2).
2. Subjects with Screening or Check-in clinical laboratory results that are outside the laboratory normal range, including hematology, clinical chemistry, serology, and urinalysis, that in the Investigator's judgment, is felt to be clinically relevant.
3. Subjects who, after 10 minutes supine rest, have a systolic blood pressure (BP) >144 mmHg or a diastolic BP >90 mmHg. If BP exceeds these cut points related to transient anxiety-related increases, BP may be repeated once.
4. Subjects with QTcF interval (Fridericia's correction factor) > 450 msec at Screening or pre dose on Day 1 of either study period.
5. Subjects with a history of serious mental illness that includes, but is not limited to, schizophrenia, bipolar disorder, and major depression. Subjects with a history of depression may be included if treatment did not require hospitalization, if the subject has been off anti-depressant medication for a minimum of 12 months, and if in the Investigator's judgment, the subject has been stable with no evidence of significant depression for a minimum of 12 months.
6. Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, cardiovascular, hepatic, hematologic, lymphatic, neurologic, endocrine, psychiatric, musculoskeletal, genitourinary, immunologic, dermatologic, or connective tissue diseases or disorders.
7. Subjects with a history of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated with no evidence of disease for at least 1 year prior to Screening.
8. Subjects with a pre-existing condition that interferes with normal gastrointestinal anatomy or motility, and/or hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study drug. Note that cholecystectomy is not exclusionary.
9. Subjects with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study.
10. Subjects who have undergone major surgery within 6 months prior to Screening.
11. Subjects who test positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection 1 or 2.
12. Subjects who have donated blood, had blood loss of more than 500 mL, or received transfusion of blood or plasma within 3 months prior to Screening.
13. Subjects who have a history of illicit drug abuse or alcoholism within 12 months prior to Screening.
14. Subjects who consume more than 21 units of alcohol a week (1 unit = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor).
15. Subjects with a positive screen for drugs of abuse, or urinary cotinine >200 ng/mL at Screening or at Check-in; subjects with a positive screen for alcohol at Check-in.
16. Subjects who are participating in any concurrent clinical trial of another investigational product or placebo, or have received an investigational agent within 2 months prior to Day 1 of Period 1.
17. Subjects who have used prescription drugs within 2 weeks or 5 half-lives (whichever is longer) of dosing on Day 1 of Period 1.
18. Subjects who have used over-the-counter (OTC) medication (excluding routine vitamins) within 7 days of dosing on Day 1 of Period 1, unless agreed as not clinically relevant by the Investigator and Sponsor's Medical Monitor. Note: use of acetaminophen up to doses no greater than 2 g in any 24 hour period up to 48 hours prior to study drug dosing is allowed.
19. Subjects who have used St. John's Wort within 28 days before dosing on Day 1 of Period 1.
20. Subjects who are unwilling to forgo consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, or grapefruit hybrids from 14 days prior to dosing on Day 1 of Period 1 through the Follow-up visit.
21. Subjects who are unwilling to forgo consumption of fruit juices, charbroiled meats, and vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard) from 7 days prior to dosing through discharge from the clinic in each period.
22. Subjects who have undergone strenuous activity within 72 hours prior to Day 1 in each period.
23. Subjects who are unable (e.g., food intolerance) or unwilling to consume a high-fat breakfast within 30 minutes.
24. Subjects with a propensity for sunburn or other skin conditions making them unsuitable for the current study.
25. Subjects who cannot communicate reliably with the Investigator.
26. Subjects who cannot or are unlikely to cooperate with the requirements of the study (for example, difficulty with swallowing multiple tablets of medication).
27. Subjects with any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in, or completion of, the study.

Ages: 18 Years to 56 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of AG-221 | Blood samples will be drawn prior to the single-dose administration of AG-221 (within 30 minutes) on Day 1 of each period, and at the following time points post dose: 1, 2, 3, 4, 6, 9, 12, 18, 24, 48, 96, 168, 240, 336, and 504 hours.
  Serial blood sampling at specified time points for determination of plasma concentration-time profiles and PK parameters of AG-221.
Incidence of adverse events | 105 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Agresta, MD, MPH &TM, Study Director — Agios Pharmaceuticals, Inc.
Locations (1):
- Baltimore, Maryland, United States